CLINICAL TRIAL: NCT05100147
Title: Comparison of Uterine Closure Techniques During Cesarean Section With Respect to the Development of Cesarean Scar Defects a Randomized Trial.
Brief Title: Uterine Closure Techniques and Cesarean Scar Defect Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Hakan Aytan, Prof. Dr. Hakan Aytan, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 473
Record Dates: First submitted 2021-10-15; First posted 2021-10-29 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Cesarean Section Complications; Scar; Deformity
Keywords: cesarean scar defect; cesarean section; uterine closure techniques
MeSH Terms: conditions — Cicatrix; Congenital Abnormalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): The uterotomy suture technique is continous, double layer suturing, in which the first layer is continuous and unlocked involving all uterine layers and a second, continuous non-locking imbrictating layer is applied over the first suture.
  Interventions: Procedure: Uterine closure during Cesarean section
- Group 2 (Experimental): The uterotomy suture technique is continous, double layer suturing, in which the first layer is continuous and unlocked not including decidua and a second, continuous non-locking imbrictating layer is applied over the first suture.
  Interventions: Procedure: Uterine closure during Cesarean section
- Group 3 (Experimental): The uterotomy suture technique is continous ,double layer with the first layer unlocked, excluding the decidua and including the deep part of the myometrium, and the second layer unlocked including the remaining part of the myometrium.
  Interventions: Procedure: Uterine closure during Cesarean section

INTERVENTIONS:
Procedure: Uterine closure during Cesarean section — The uterotomy is sutured after the delivery of the fetus and the placenta with an appropriate delayed absorbable suture (number 1 polyglactin 910)

SUMMARY:
Cesarean operations are one of the most common obsetric operations and have an increasing trend in all over the world. However unfortunately the operation techniques have not been standardized yet. It is well known that different uterine closure techniques result in differences with respect to wound healing on the uterus; however, the ideal uterine closure technique is yet not known. The aim of this study is to assess the results of different uterine closure techniques during cesarean section with respect to the development of cesarean scar defects.

DETAILED DESCRIPTION:
Patients were randomized into three groups using a computer-based program (ratio 1:1:1), and the assigned surgical technique was disclosed just before surgery. At the time of surgery, the sealed opaque envelope, numbered consecutively and containing the description of the suturation technique, was given to the operator. Suturing techniques varied between groups: double layer continuous, non-locking suturing with endometrial inclusion, second layer imbricating the first layer (Group 1), double layer, continuous, non-locking suturing without endometrial inclusion second layer imbricating the first layer (Group 2) and double layer continuous with the first layer unlocked, including the endometrium and the deep part of the myometrium, and the second layer continuous unlocked including the remaining part of the myometrium (Group 3) (Figure 2). Size 1 polyglycolic acid 910 (Vicryl ® Ethicon Inc. Somerville, NJ) was used as suture material in all groups.

Patients were re-evaluated at the sixth month as uterine scar healing is reported to be completed within six months and preoperative assessments were repeated. Transvaginal ultrasonography was performed by an investigator blinded to suturing techniques. Measurements included RMT, and CSD assessment (as the primary outcomes) (including the depth and width of the CSD), as well as other routine ultrasonographic evaluations. Transvaginal sonography was performed by the same investigator with a Toshiba Applio 500 device using a PMW-621VT 6 Mhz R13 probe. CSD was considered when myometrial continuity in the previous caesarean incision site was lost, and an anechoic defective area towards the myometrium was noted. In patients who did not develop CSD, the incision line was measured anteriorly, and the symmetrical posterior uterine wall thickness was measured. In patients with CSD, the myometrium tissue above the anechoic defective area was evaluated as residual myometrial thickness. The CSD sac's depth and its base's width were measured. The full-thickness myometrium adjacent to the defect area was measured, and recovery rates were calculated by taking the percentage of the residual myometrial thickness over the defect to the full-thickness myometrium.

ELIGIBILITY:
Inclusion Criteria:

1. being nulliparous
2. having singleton fetus
3. not having diabetes and or hypertension
4. not having an intrauterine infection
5. body mass index <35 kg/m2
6. not having any placental insertion anomalies
7. not having Mullerian anomalies
8. active phase of labor is not started.
9. no previous uterine surgeries

Exclusion Criteria:

1. being multiparous
2. having multiple pregnancies
3. having diabetes and or hypertension
4. having an intrauterine infection
5. body mass index >=35 kg/m2
6. having any placental insertion anomalies
7. having Mullerian anomalies
8. in active phase of labor
9. having previous uterine surgeries

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Scar thickness at postpartum 6th week | Postpartum 6th weeks
  The patients will be examined at the postpartum sixth week. During that visit uterine scar thickness will be measured by ultrasound. Measurement of uterine scar thickness will be performed perpendicular to the uterine wall and calipers will be placed on the serosal surface of the uterus and the delineation of the endometrium. These landmarks represent the inner and outer edge of the Cesarean scar.
Scar thickness at postpartum 6th month | Postpartum 6th months
  The patients will be reexamined at the postpartum sixth month. During that visit uterine scar thickness will be measured again. Measurement of uterine scar thickness will be performed with the same method (perpendicular to the uterine wall and calipers will be placed on the serosal surface of the uterus and the delineation of the endometrium. These landmarks represent the inner and outer edge of the Cesarean scar.)

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Oktay, MD, Study Chair — Mersin University Hospital
Locations (1):
- Mersin University Hospital, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No